CLINICAL TRIAL: NCT05071235
Title: Quality of Life of Patients With Diabetic Foot Ulcers Treated With LLLT 904 nm and Aspects Associated With Self-care Adherence: a Randomized Clinical Trial
Brief Title: Quality of Life and Self-care in Patients With Diabetic Foot Ulcers Treated With Low-level Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Vinicius Saura Cardoso, PhD Professor of the Graduate Program in Biomedical Sciences, Federal University of Piaui
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3.533.413
Record Dates: First submitted 2021-09-13; First posted 2021-10-08 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Control Groups; Bandages

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CG (control group) + dressing (Placebo Comparator): The group will receive placebo LLLT (low-level laser therapy) application associated with Helianthus annuus oil dressing.
  Interventions: Device: CG (control group); Procedure: Dressing
- LG1 (LLLT group 1) + dressing (Active Comparator): The group will receive application of LLLT (low-level laser therapy) Gallium Arsenide (GaAs) 904 nm 10 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: LG1 (LLLT group 1); Procedure: Dressing
- LG2 (LLLT group 2) + dressing (Active Comparator): The group will receive application of LLLT (low-level laser therapy) Gallium Arsenide (GaAs) 904 nm 8 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: LG2 (LLLT group 2); Procedure: Dressing
- LG3 (LLLT group 3) + dressing (Active Comparator): The group will receive application of LLLT (low-level laser therapy) Gallium Arsenide (GaAs) 904 nm 4 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: LG3 (LLLT group 3); Procedure: Dressing

INTERVENTIONS:
Device: LG1 (LLLT group 1) — Application of LLLT (low-level laser therapy) AsGa 904 nm 10 J/cm².
  Arms: LG1 (LLLT group 1) + dressing
Device: LG2 (LLLT group 2) — Application of LLLT (low-level laser therapy) AsGa 904 nm 8 J/cm².
  Arms: LG2 (LLLT group 2) + dressing
Device: LG3 (LLLT group 3) — Application of LLLT (low-level laser therapy) AsGa 904 nm 4 J/cm².
  Arms: LG3 (LLLT group 3) + dressing
Device: CG (control group) — Application of placebo LLLT (low-level laser therapy), that is, with the device turned off.
  Arms: CG (control group) + dressing
Procedure: Dressing — Application of Helianthus annuus oil dressing.

SUMMARY:
Diabetic foot ulcers (DFU) are aggressive complications of diabetes mellitus (DM) and affect 25% of these patients. DFU are associated with a high risk of amputations and early mortality and significantly impact quality of life (QoL). The low-level laser therapy (LLLT) is an important approach for the treatment of DFU, however there is a lack of data on its influence on the QoL of patients with DFU. On the other hand, adherence to self-care is a factor closely related to QoL. Therefore, this study is justified by the need to understand the impact of LLLT on QoL and its relationship with self-care. Aim: To evaluate the quality of life of patients with diabetic foot ulcers treated with different doses of LLLT (GaAs) 904 nm and its association with aspects of adherence to self-care. Methods: This is a randomized, double-blind, placebo-controlled clinical trial. Participants will be randomly assigned to the groups: control LLLT placebo (CG), LLLT 904 nm 10 J/cm² (LG1), LLLT 904 nm 8 J/cm² (LG2) and LLLT 904 nm 4 J/cm² (LG3). QoL data, percentage of healing and pain will be assessed before the start of the intervention, in 10th week and after one month to the end of intervention, self-care will be assessed before the start of the intervention and at the end of intervention. Eighty participants with DFU will be recruited who will receive intervention twice a week for up to 20 visits (10 weeks).

DETAILED DESCRIPTION:
Eighty volunteers will be recruited through the Integrated Center of Medical Specialties (ICMS) and the Center of Health Specialties (CHS) in Parnaíba-PI, Brazil, after thorough examination of the feet and evaluation by a medical professional specializing in vascular surgery. Volunteers with type 2 diabetes mellitus (T2DM) who have DFU without an infectious process (Wagner's grade I and II) will be admitted, of both sexes aged 18 years and over. Inclusion in the study will take place after signing the Informed Consent Form (ICF). The randomization will be of the simple type, a computer generated randomization list through the website https://www.randomizer.org will be used to prepare sealed, opaque and sequentially numbered envelopes. A collaborator, who will not participate in the study, will carry out the randomization process, subsequently inserting the allocation data in the envelope.

After inclusion, volunteers will be evaluated individually in a reserved room, by a previously trained evaluator and blinded to the allocation of volunteers in the groups. Volunteers will provide their personal data, medical history and duration of T2DM. Subsequently, the physical evaluation and application of the questionnaires will be carried out: (1) application of the SF-36 (Short Form-36 Health Survey) and Summary of Diabetes Self-Care Activities (SDSCA) questionnaires in the form of an interview; (2) vascular evaluation; (3) neurological evaluation; (4) determination of the level of pain and (5) capillary blood glucose.

The DFU will be located, recording the affected foot region, the duration in months and the Wagner's classification. The healing process of DFU will be monitored. The total number of LLLT applications performed until complete healing will be identified and the percentage of patients who achieved healing in relation to the cutoff points of the fifth and tenth weeks of intervention. The volunteers in the treatment groups will receive dosage as pre-established (10, 8 or 4 J/cm²) and those in the control group (CG) will receive a placebo application, that is, with the device turned off. For the treatment, the laser tip will be positioned perpendicular to the DFU, the ulcer floor will be irradiated with a sweeping application technique (1 cm away from the ulcer) and the edges with a punctual technique with contact at equidistant points. The total duration of each application will be calculated by the machine based on the selected energy density. Both the therapist and the participant will use the goggles provided before the application. The four groups will receive conventional treatment, cleansing the ulcers with saline solution and dressing with Helianthus Annuus oil.

It is expected that the participants in the treatment groups will show significant improvement in QoL and pain after the intervention, less time and a higher percentage of healing compared to the CG. Differences in the improvement of QoL and pain and in the time and percentage of healing between the LLLT dosages used are also expected. It is also assumed that adherence to self-care is capable of predicting the time and percentage of healing and QoL, in the perception that the improvement of the patient with LLLT is also influenced by his attitudes and that self-care also has effects on QoL.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients with diabetic foot ulcers;
* Patients aged 18 to 79 years.

Exclusion Criteria:

* Presence of autoimmune disease;
* Presence of psychiatric or cognitive disorders that impede the application of questionnaires;
* Pressure ulcers
* Venous ulcers;
* Contraindications to the treatment methods adopted in the research;
* Ulcers in other parts of the body than the feet;
* Diabetic foot ulcers infected.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Initial quality of life (QoL) | Before intervention starts.
  Quality of life assessed by the SF-36 questionnaire.
Final quality of life (QoL) | In 10th week of intervention or after DFU healing (in ulcers that healed before 10 weeks).
  Quality of life assessed by the SF-36 questionnaire.
Quality of life (QoL) follow up | 1 month after the end of the intervention.
  Quality of life assessed by the SF-36 questionnaire.

SECONDARY OUTCOMES:
Healing time | In 10th week of intervention or after DFU healing (in ulcers that healed before 10 weeks).
  Total applications performed until healing.
Percentage of complete healing in 5th week | In 5th week of intervention.
  Percentage of patients achieving healing in each group.
Percentage of complete healing in 10th week | In 10th week of intervention.
  Percentage of patients achieving healing in each group.
Percentage of complete healing follow up | 1 month after the end of the final intervention.
  Percentage of patients achieving healing in each group.
Self-care | Before intervention starts.
  Adherence to self-care assessed by the Summary of Diabetes Self-Care Activities (SDSCA) questionnaire.
Change in self-care | In 10th week of intervention or after DFU healing (in ulcers that healed before 10 weeks).
  Adherence to self-care assessed by the Summary of Diabetes Self-Care Activities (SDSCA) questionnaire.
Visual analogue scale (VAS) | Before intervention starts.
  Levels of pain in the feet assessed using the visual analogue scale (VAS). With scores ranging from 0 to 100, 0 being no pain and 100 being the worst pain that the patient imagines.
Change in visual analogue scale (VAS) | In 10th week of intervention or after DFU healing (in ulcers that healed before 10 weeks).
  Levels of pain in the feet assessed using the visual analogue scale (VAS). With scores ranging from 0 to 100, 0 being no pain and 100 being the worst pain that the patient imagines.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Piaui, Parnaíba, Piauí, Brazil